CLINICAL TRIAL: NCT02117492
Title: A Randomized Trial Comparing Horizontal and Vertical Vaginal Cuff Closure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Timothy A Deimling, Minimally Invastive GYN Surgery, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 00000143
Record Dates: First submitted 2014-04-16; First posted 2014-04-21 (Estimated); Last update posted 2017-09-20 (Actual); Status verified 2017-09

CONDITIONS: Hysterectomy
Keywords: hysterectomy; vaginal cuff

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vertical Cuff (Experimental): Vaginal cuff closure will be done vertically.
  Interventions: Procedure: Cuff Closure
- Horizontal Cuff (Experimental): Vaginal cuff closure will be done horizontally.
  Interventions: Procedure: Cuff Closure

INTERVENTIONS:
Procedure: Cuff Closure — Closure of the vaginal cuff following hysterectomy.

SUMMARY:
The purpose of this study is to evaluate the possible impacts of two techniques of vaginal cuff closure during robotic hysterectomy. We aim to compare vertical vs horizontal vaginal cuff closure and the impact that these techniques have on vaginal length, sexual function, and overall complication rates.

DETAILED DESCRIPTION:
A Validated questionnaire the Female Sexual Function Index (FSFI) and total vaginal lengths will be used to evaluate patients pre-operatively, at 4-6 weeks post-operatively, and 6 months post operatively. The FSFI will also be sent to the patient 12 months post operatively. These data will be used to assess sexual function and total vaginal length in patients undergoing minimally invasive hysterectomy. The study endpoint will occur after the 12 month follow-up questionnaire. Additionally, all complications following surgery will be tracked over the study period for comparison.

ELIGIBILITY:
Inclusion Criteria:

1. Female premenopausal patients undergoing robot assisted total laparoscopic hysterectomy

Exclusion Criteria:

1. Adults unable to consent
2. Children under the age of 18
3. Pregnant women
4. Prisoners
5. Post-menopausal women
6. Women with the known preoperative need for bowel or genitourinary surgery at the time of hysterectomy
7. Patients unable to consent to the procedure in the English language

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Vaginal Length | up to 4-6 weeks post-operative
  The primary endpoint measured in the study will be total vaginal length. This will be measured preoperatively, at 4-6 weeks postoperatively.

SECONDARY OUTCOMES:
Sexual Function | Pre-operative, 6 and 12 months post-operativey
  Secondary outcomes will include sexual function measured with FSFI preoperatively and at 6 months and 12 months post operatively.

OTHER OUTCOMES:
Complication Rates | up to 12 months post-operativey
  Overall complication rates will be monitored.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy A Deimling, MD, MS, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Penn State Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No